CLINICAL TRIAL: NCT06805812
Title: Predictive Impact of Peripheral Blood Lymphocytes on clinicAL outcoMes During First-line CDK4/6 Inhibitors Plus Endocrine Therapy in Patients With Advanced Hormone REceptor-poSitive HER2-negative Breast Cancer: the Retrospective-prospective Multicenter Italian PALMARES-2 Study
Brief Title: Predicting clinicAL outcoMes During First-line CDK4/6 Inhibitors Plus Endocrine Therapy in Patients With Advanced Hormone REceptor-poSitive HER2-negative Breast Cancer: the Retrospective-prospective Multicenter Italian PALMARES-2 Study
Acronym: PALMARES-2
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: European Institute of Oncology, Italy (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); OSPEDALE ASST CREMONA (Unknown); IOV Oncologico Veneto Padova (Unknown); ASST Fatebenefratelli Sacco (Other); IRCCS Fondazione Salvatore Maugeri, Pavia, Italy (Unknown); IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori Meldola (Unknown); Azienda Ospedaliero-Universitaria di Modena (Other); Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara (Unknown); A.O.U. Federico II, Napoli (Unknown); San Raffaele University Hospital, Italy (Other); Centro di Riferimento Oncologico - Aviano (Other); Azienda Socio-Sanitaria Territoriale Lariana (Unknown); Azienda ULSS 3 Serenissima, Ospedale di Mirano (Unknown); Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma (Unknown); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Humanitas, Istituto Clinico Catanese (Other Government); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Fondazione Policlinico Universitario Campus Bio-Medico (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: INT101/23
Record Dates: First submitted 2025-01-07; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Breast Adenocarcinoma; Breast Cancer Stage IV; Breast Cancer, Metastatic; Breast Carcinoma; Breast Diseases; Breast Neoplasms; Breast Neoplasms, Male; Breast Cancer; Breast Cancer With Metastatic Bone Disease; Breast Cancers; Breast Neoplasm; Breast Tumors; HR+ HER2- Men, Pre/Postmenopausal Advanced Breast Cancer; HR+ Advanced or Metastatic Breast Cancer; HR+/HER2- Breast Cancer; HRpos Breast Neoplasms; HR-positive, HER2-negative Advanced Breast Cancer; HR-positive, HER2-negative and PIK3CA Mutation Advanced Breast Cancer; HR-positive Breast Cancer; Hormone Receptor-Positive Breast Cancer; Hormone Receptor Positive Breast Adenocarcinoma; Hormone Receptor Positive Breast Carcinoma; Hormone Receptor Positive Breast Neoplasms; Hormone Receptor Positive HER-2 Negative Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast; Hormone Receptor Positive Metastatic Breast Cancer; Hormone Receptor Positive, HER2 Negative Breast Cancer; Hormone Receptor Negative Breast Cancer; Hormone Receptor Positive, HER2-negative, Advanced Breast Cancer; Hormone Receptor Positive Breast Cancer; Hormone Receptor Positive (ER+/PR+, and Her2-) Metastatic Breast Cancer; Hormone Receptor Positive, HER2-negative Neoplasms; Hormone Receptor Positive, HER2-low Neoplasms; Hormone Receptor Positive (HR+), HER2-negative Breast Cancer; Hormone Receptor (HR)-Positive Breast Cancer; Hormone Receptor-Positive, HER2-Negative Metastatic Breast Cancer; Palbociclib; Ribociclib; Abemaciclib; CDK4/6 Inhibitor; CDK4/6 Inhibitors
Keywords: HR+/HER2- Advanced Breast Cancer; HR+/HER2- Metastatic Breast Cancer; Palbociclib; Ribociclib; Abemaciclib; CDK4/6i; Cyclin-Dependent Kinase 4/6 inhibitors; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Breast Diseases; Breast Neoplasms, Male | interventions — palbociclib; ribociclib; abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Archival tumor FFPE block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Palbociclib — Administered in combination with endocrine therapy
Drug: Ribociclib — Administered in combination with endocrine therapy
Drug: Abemaciclib — Administered in combination with endocrine therapy

SUMMARY:
PALMARES-2 is a retrospective/prospective, observational, multicenter, population-based study, aiming at providing real-world evidences on HR+/HER2- aBC patients treated with first-line CDK4/6i plus ET. The present study has the objective to collect data coming from different sources, i.e. RWD, medical images and biological samples, from patients treated with CDK4/6i as first-line of therapy for HR+/HER2- aBC. In consideration of the complexity of data collected and different objectives of the study, this master protocol foresees different sub-studies, which encompasses different methodologies for data collection, data extraction and analyses.

DETAILED DESCRIPTION:
The PALMARES-2 study aims to collect data from different sources, i.e. real-world clinical data, medical images and biological data and samples, from patients treated with CDK4/6i as first-line therapy for patients with HR+/HER2- advanced breast cancer. Due to the complexity of the data collected and the different objectives of the study, this protocol includes several sub-studies, which include different methodologies for data collection, extraction and analysis:

* The first sub-study (RWD sub-study) will aim to collect real-world clinical data of patients who received ET+CDK4/6i in the first-line setting; the primary objective of this sub-study is to assess whether there is a difference in OS between the three CDK4/6i in the real-world population, while secondary objectives include comparisons in specific sub-groups;
* The second sub-study (Safety sub-study) includes the collection of comorbidities, concomitant medications and toxicities of patients enrolled in the study; the primary objective of this sub-study is to evaluate the difference in severe toxicity between the three CDK4/6i in the real-world population
* The third sub-study (medical imaging sub-study) consists of the collection of computed tomography (CT) and fluorodeoxyglucose positron emission tomography (FdG-PET) images at baseline and digitised haematoxylin-eosin (HE) slides to build a multi-omics predictive model;
* The fourth sub-study (translational sub-study) aims to collect tumour samples from a proportion of patients enrolled in the study to perform genomics and transcriptomics analyses; information from this data source will be integrated into the model built with the previous data to further improve the performance of the previous model
* The fifth sub-study (subsequent lines sub-study) focuses on the lines of treatment administered to patients enrolled in the study at the time of progression after first-line treatment with ET+CDK4/6i, with the aim of building predictive models of response to subsequent lines of treatment, capable of supporting oncologists' and patients' decisions in this context.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HR+/HER2- advanced Breast Cancer (aBC), as defined as at least 1% estrogen receptor (ER) and/or progesterone receptor (PgR) positivity at IHC. HER2 negativity is defined on the basis of an IHC score of 0, 1+, or 2+ with absence of gene amplification at in situ hybridization (ISH) analyses.
* Have received or are candidate to receive treatment with palbociclib, ribociclib or abemaciclib in combination with endocrine therapy as first-line treatment for HR+/HER2- aBC.

Exclusion Criteria:

* Less than 3 months of follow up from the CDK4/6i start to the date of data cut-off;
* Have received CDK4/6i as monotherapy;
* Have received CDK4/6i as adjuvant treatment for localized disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the retrospective and prospective collection of consecutive HR+/HER2- advanced Breast Cancer patients (defined as metastatic or locally advanced not candidate for definitive curative intervention) treated with CDK4/6i in combination with endocrine therapy as first-line treatment for advanced disease in different Italian cancer centers.
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the first-line treatment start to date of any-cause death or last follow up, up to 120 months

SECONDARY OUTCOMES:
Real-world Progression-Free Survival (rwPFS) | From the start of first-line treatment to date of disease progression documented in patient medical charts or death or last follow up, whichever occurs first, up to 120 months
Time To Next Treatment or Death (TTNT-D) | From the start of first-line treatment to date of subsequent therapy start or death or last follow up, whichever occurs first, up to 120 months
Time To Chemotherapy or Death (TTC-D) | From the start of first-line treatment to date of first chemotherapy for advanced disease start or death or last follow up, whichever occurs first, up to 120 months

CONTACTS AND LOCATIONS:
Locations (24):
- Italy (24):
  - Centro di Riferimento Oncologico IRCCS, Aviano
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili, Brescia
  - Humanitas Istituto Clinico Catanese, Catania
  - ASST Lariana - Ospedale Sant'Anna, Como
  - ASST Ospedale Maggiore, Cremona
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Istituto Tumori della Romagna IRST IRCCS, Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale ASST Fatebenefratelli Sacco, Milan
  - ULSS 3 Veneto, Mirano
  - Azienda Ospedaliero-Universitaria, Modena
  - Azienda Ospedaliero-Universitaria Federico II, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Ospedale Maggiore della Carità, Novara
  - IOV Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS - ICS Maugeri, Pavia
  - Clinica Ospedaliero - Universitaria Policlinico Umberto I, Roma
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be evaluated for submission

DOCUMENTS (1):
  • Study Protocol (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT06805812/Prot_000.pdf